CLINICAL TRIAL: NCT01363336
Title: Post-marketing Surveillance for Hypertensive Patients With Diabetes and/or Chronic Kidney Disease
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 15190
Record Dates: First submitted 2011-04-28; First posted 2011-06-01 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2015-04

CONDITIONS: Hypertension
Keywords: Adalat; Hypertension; Diabetes; Chronic kidney disease
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Renal Insufficiency, Chronic | interventions — Nifedipine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Nifedipine (Adalat CR, BAYA1040)

INTERVENTIONS:
Drug: Nifedipine (Adalat CR, BAYA1040) — patients who are administrated with Adalat CR for hypertension

SUMMARY:
This study is a post-marketing surveillance in Japan, and it is a local prospective, company sponsored and observational study of patient who have been treated by Adalat CR for hypertension with diabetes and/or chronic kidney disease. The objective of this study is to assess safety and efficacy profile of using Adalat CR in real clinical practice. A total 2,000 patients will be recruited and be observed for 6 months. Then, patient of whom microalbumin urea and serum creatinine are continuously monitored are additionally followed for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient who are administered with Adalat CR for hypertension with diabetes and/or chronic kidney disease (CKD)

Exclusion Criteria:

* CKD with stage 5
* CDK with dialysis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The target population of this study is patient who have been administered with Adalat CR for hypertension with diabetes and/or chronic kidney disease. The study is expected to collect data of 2,000 pateints in Japan.
Sampling Method: Non-Probability Sample
Enrollment: 1882 (Actual)
Dates: Start 2009-11; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of participants with Adverse Events for Safety purpose in real practice | After 6 months
General evaluation of patient concerning efficacy of AdalatCR treatment in real practice | After 6 months

SECONDARY OUTCOMES:
Blood pressure, Pulse rate | After 6 months
Clinical test values, in specially, microalbumin urea and serum creatinine | After 6 months
Overall evaluation | After 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Japan